CLINICAL TRIAL: NCT02815813
Title: Peer Support and Mobile Technology Targeting Cardiometabolic Risk Reduction in Young Adults With Serious Mental Illness
Brief Title: Lifestyle Intervention for Young Adults With Serious Mental Illness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Kelly Aschbrenner, PhD, Senior Scientist, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STUDY00029586; R01MH110965 (NIH)
Record Dates: First submitted 2016-06-24; First posted 2016-06-28 (Estimated); Results first posted 2025-01-14 (Actual); Last update posted 2025-01-14 (Actual); Status verified 2024-11

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Bipolar Disorder; Major Depressive Disorder; Overweight; Obesity
Keywords: Serious Mental Illness; Young Adults; Obesity; Cardiometabolic Risk; Physical Activity; Weight Loss; Fitness; Peer Support; Smartphone; Mobile Technology; mHealth; Social Media; Facebook; Lifestyle Intervention
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Bipolar Disorder; Depressive Disorder, Major; Overweight; Obesity; Motor Activity; Weight Loss

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PeerFIT (Experimental): PeerFIT is a group-based lifestyle intervention enhanced by mobile health technology and social media designed to achieve clinically significant improvements in weight loss and cardiorespiratory fitness in young adults with serious mental illness.
  Interventions: Behavioral: PeerFIT
- BEAT (Active Comparator): BEAT involves basic education in fitness and nutrition supported by a wearable activity tracking device designed to achieve clinically significant improvements in weight loss and cardiorespiratory fitness in young adults with serious mental illness.
  Interventions: Behavioral: BEAT

INTERVENTIONS:
Behavioral: PeerFIT — The 12-month PeerFIT intervention consists of a 6-month intensive phase including: (a) once weekly 60-minute group weight management and exercise session led by a lifestyle coach; (b) once weekly one-hour physical activity session delivered in community settings; and (c) Facebook and mHealth technology (i.e., Fitbits, text messaging support) to increase motivation and facilitate self-monitoring and peer social support for health behavior change. Participants then transition to a 6-month lower intensity phase in which the 90-minute weight management sessions are discontinued. The groups will be conducted as open groups with a minimum of 4 and maximum of 18 participants at any given time.
  Arms: PeerFIT
Behavioral: BEAT — Participants in BEAT will receive monthly individual lifestyle sessions delivered by a lifestyle coach including education, guidance, and support for self-monitoring behaviors (i.e., daily self-weighing and tracking daily steps) during the first six months of the study, plus text message reminders and encouragement for self-monitoring weight loss behaviors during the entire 12-month study period. Participants will receive materials with tips and strategies for healthy eating and increasing physical activity. They will also be given a wearable activity tracker (i.e., Fitbit Zip) to use with instructions for using the device. The first session with the lifestyle coach will be in person and thereafter by phone.
  Arms: BEAT

SUMMARY:
This is a four year project evaluating the effectiveness of a group-based lifestyle intervention (PeerFIT) supported by mobile health (mHealth) technology and social media compared to Basic Education in fitness and nutrition supported by a wearable Activity Tracking device (BEAT) in achieving clinically significant improvements in weight loss and cardiorespiratory fitness in young adults with serious mental illness (SMI).

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effectiveness of a group-based lifestyle intervention (PeerFIT) supported by mobile health (mHealth) technology and social media to promote weight loss and improved fitness in young adults with serious mental illness (SMI). The study is a two-arm randomized controlled trial conducted in real world mental health settings to evaluate the effectiveness of the 12-month PeerFIT intervention compared to Basic Education in fitness and nutrition supported by a wearable Activity Tracking device (BEAT) in achieving clinically significant improvements in weight loss and cardiorespiratory fitness. The investigators will enroll 144 overweight and obese (BMI ≥ 25) young adults ages 18 to 35 with SMI attending one of two community mental health who are interested in losing weight and improving fitness. The investigators hypothesize that PeerFIT compared to BEAT will be associated with a greater proportion of participants who achieve cardiovascular risk reduction at 6 and 12 months follow-up as indicated by either clinically significant weight loss (5% or greater) or increased fitness (>50 m on the six-minute walk test). The investigators also hypothesize that PeerFIT compared to BEAT will be associated with greater improvements in A1c and lipid profiles at 6 and 12 months follow-up. They will also investigate two theoretical mechanisms of action hypothesized to account for greater weight loss and increased cardiorespiratory fitness among participants assigned to PeerFIT: 1) improved self-efficacy and 2) increased peer support for health behavior change. The investigators hypothesize that the relationship between PeerFIT and weight loss and improved fitness will be mediated by improved self-efficacy and peer support for health behavior change.

ELIGIBILITY:
Inclusion Criteria:

* Young adults ages 18 to 35
* Chart diagnosis of schizophrenia, schizoaffective disorder, bipolar disorder, or major depression
* Overweight or obese defined as BMI ≥25
* Enrolled in treatment at the agency for at least 3 months prior to study recruitment
* Have not started taking Clozapine or Olanzapine antipsychotic medications over the prior 2 months (dose changes are allowed)
* Able and willing to give written informed consent to participate in the study or able to assent with guardian consent
* Willingness to be randomized to either of the two conditions
* Able and willing to attend the weekly 60-minute weight management session, participate in the weekly 1-hour physical activity sessions, and use the Facebook and mHealth (i.e., Fitbits and text messaging) components of the PeerFIT program

Exclusion Criteria:

* Medical contraindication to weight loss (e.g., cancer, stroke, liver failure)
* Medical conditions (e.g., diabetes, angina) that do not receive medical clearance by a primary care provider
* Major surgery planned or likely to occur within the next 6 months
* Prior or planned bariatric surgery
* Use of prescription weight loss medication within the past 6 months
* 5% or greater weight loss in 3 months prior to baseline
* Currently enrolled in another weight reduction program
* Pregnant or planning a pregnancy, or breastfeeding during study period
* Cognitive impairment sufficient to interfere with participant's ability to provide informed consent, complete study questionnaires, or participate in a group intervention as indicated by a Mini Mental Status Examination score <24
* Active substance use determined to be incompatible with participation in the intervention identified by screening questionnaire that assesses for excessive use according to intake limits by gender
* Use of anabolic steroids with the drug taken at least "most days of the week for the previous month"
* Planning to leave agency or move out of geographic area within 12 months
* People who are non-English speakers or who have major visual or hearing impairment will be excluded given the need to read the program materials and interact with technology.

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 150 (Actual)
Dates: Start 2017-07-03 (Actual); Primary Completion 2022-05-31 (Actual); Study Completion 2022-05-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelly A Aschbrenner, PhD, Principal Investigator — Dartmouth-Hitchcock and Geisel School of Medicine at Dartmouth College
Locations (2):
- United States (2):
  - Community Mental Health Affiliates, New Britain, Connecticut
  - Greater Nashua Mental Health Center, Nashua, New Hampshire

IPD SHARING:
Plan to Share IPD: Yes
The proposed project involves human subject data, and all data collected on subjects (both positive and negative) will be submitted to the National Database for Clinical Trials Related to Mental Illness (NDCT). This will include individual level data from all subjects enrolled in both the active intervention and control conditions.
  The NDCT is a secure data repository run by the National Institute of Mental Health (NIMH) that allows researchers to collect and share de-identified information with each other. This secure informatics platform facilitates scientific collaboration and data sharing, and enables effective communication of detailed research data, tools, and supporting documentation. The NDCT links data across research projects using Global Unique Identifiers (GUID) for each participant, and the NDCT Data Dictionary.

REFERENCES:
- [Derived] Aschbrenner KA, Naslund JA, Gorin AA, Mueser KT, Browne J, Wolfe RS, Xie H, Bartels SJ. Group Lifestyle Intervention With Mobile Health for Young Adults With Serious Mental Illness: A Randomized Controlled Trial. Psychiatr Serv. 2022 Feb 1;73(2):141-148. doi: 10.1176/appi.ps.202100047. Epub 2021 Jun 30. PMID 34189933
- [Derived] Aschbrenner KA, Naslund JA, Gorin AA, Mueser KT, Scherer EA, Viron M, Kinney A, Bartels SJ. Peer support and mobile health technology targeting obesity-related cardiovascular risk in young adults with serious mental illness: Protocol for a randomized controlled trial. Contemp Clin Trials. 2018 Nov;74:97-106. doi: 10.1016/j.cct.2018.10.005. Epub 2018 Oct 11. PMID 30316998

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | PeerFIT | BEAT
Started | 76 | 74
Completed | 53 | 51
Not Completed | 23 | 23

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | PeerFIT | BEAT | Total
Number analyzed (Participants) | 76 | 74 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.2 (4.4) | 28.5 (4.7) | 28.4 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 41 | 42 | 83
  Male | 35 | 32 | 67
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 23 | 45
  Not Hispanic or Latino | 54 | 51 | 105
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 1 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 18 | 21 | 39
  White | 44 | 38 | 82
  More than one race | 6 | 6 | 12
  Unknown or Not Reported | 7 | 9 | 16
Region of Enrollment [Number; unit: participants] — All participants in this study were enrolled from clinic sites located in the U.S.
  participants
    United States | 76 | 74 | 150

OUTCOME MEASURES:

1. Primary Outcome: Weight
Description: Participants' weight will be measured in pounds (lbs.) on a flat, even surface with the use of a high-quality, calibrated professional medical scale, with the participant wearing indoor clothing and no shoes.
Time Frame: Baseline, 6 months, and 12 months
Population: Participants at baseline, 6 months and 12 months
Measure: Mean (Standard Deviation); unit: Kilogram
Arm/Group | PeerFIT | BEAT
Number analyzed (Participants) | 76 | 74
Kilogram
  Baseline weight | 107.6 (26.9) | 105.1 (20.9)
  6-month weight | 109.7 (26.3) | 106.7 (22.1)
  12-month weight | 109.2 (27.6) | 106.9 (22.5)
Statistical Analysis 1: Comparison: PeerFIT vs BEAT; Test type: Superiority; p < 0.01, GLMM

2. Primary Outcome: 6-minute Walk Test
Description: After a baseline blood pressure has been obtained, participants are asked to walk a measured distance as far as they are able in 6 minutes.
Time Frame: Baseline, 6 months, and 12 months
Measure: Mean (Standard Deviation); unit: feet
Arm/Group | PeerFIT | BEAT
Number analyzed (Participants) | 76 | 74
feet
  Baseline | 1398 (296) | 1424 (250)
  6-months | 1386 (296) | 1426 (248)
  12-months | 1357 (271) | 1319 (332)
Statistical Analysis 1: Comparison: PeerFIT vs BEAT; Test type: Superiority; p < 0.01, GLMM

3. Secondary Outcome: Self-efficacy for Exercise Behaviors Assessed Using the Self-efficacy for Exercise Behaviors (SEB) Scale
Description: The Self-efficacy for Exercise Behaviors (SEB) scale was used to measure participants' self-efficacy related to the ability to exercise despite common barriers. Five items represent the following areas:
  negative affect, resisting relapse, and making time for exercise. Respondents rate their confidence on a five-point Likert scale from 1 = "I know I cannot" to 4 = "I know I can". Total scores range from 5 to 20. Higher overall scores indicate higher exercise self efficacy.
Time Frame: Six months and 12 months
Population: Data analyzed at 6 months for both PeerFIT and BEAT arms.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PeerFIT | BEAT
Number analyzed (Participants) | 54 | 49
score on a scale
  6 months | 11 (3.4) | 10.7 (4.3)
  12 months: number analyzed (Participants) | 45 | 43
  12 months | 11.2 (3.5) | 10.2 (3.4)

4. Secondary Outcome: Social Provisions Scale (SPS)
Description: Participants' level of perceived peer support was measured with the Social Provisions Scale (SPS). The SPS consists of 10 questions items assessing an individual's perceived social support across different dimensions like attachment, guidance, social integration, reliable alliance, and reassurance of worth; essentially assessing how much support they feel they receive from their social network. The items are rated on a 4-point Likert scale from 1 ("strongly disagree) to 4 ("strongly agree") as it pertains to relationships with group members. Scores range from 10 to 40. Higher scores indicate greater perceived support from group relationships.
Time Frame: Six months and 12 months
Population: Data was collected on SPS for the PeerFIT group only at 6 and 12 months.
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | PeerFIT
Number analyzed (Participants) | 47
score on a scale
  6 months | 29.2 (5.2)
  12 months: number analyzed (Participants) | 27
  12 months | 27.1 (5.9)

5. Secondary Outcome: Hemoglobin A1C
Description: Hemoglobin A1C will be measured using the CardioChek PA Analyzer.
Time Frame: Baseline, 6 months, and 12 months
Population: Analyzed at baseline, 6 and 12 months
Measure: Mean (Standard Deviation); unit: Percentage of HbA1c
Arm/Group | PeerFIT | BEAT
Number analyzed (Participants) | 76 | 74
Percentage of HbA1c
  Baseline | 5.3 (0.8) | 5.3 (1.0)
  6 months | 5.3 (0.7) | 5.3 (0.6)
  12 months | 5.6 (1.4) | 5.5 (0.7)

ADVERSE EVENTS:
Time Frame: 1 year
Groups:
- PeerFIT: Group based lifestyle intervention
- BEAT: Remote lifestyle intervention
Arm/Group | PeerFIT | BEAT
All-Cause Mortality (participants affected / at risk) | 0/76 | 0/74
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/74
Other Adverse Events (participants affected / at risk) | 0/76 | 0/74

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-05-20): https://cdn.clinicaltrials.gov/large-docs/13/NCT02815813/Prot_SAP_000.pdf